CLINICAL TRIAL: NCT05924633
Title: A Study of a Dietary Supplement in Breastfeeding Mothers (WellFed)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Aifric O'Sullivan, Assistant Professor and Principal Investigator, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LS-23-07-OSullivan
Record Dates: First submitted 2023-06-08; First posted 2023-06-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dietary Habits; Dietary Supplements; Maternal Health; Breastfeeding; Infant Health
Keywords: Breastfeeding; Dietary Supplements
MeSH Terms: conditions — Feeding Behavior; Breast Feeding | interventions — beta-Glucans

STUDY DESIGN:
Intervention Model Description: Parallel randomised control trail
Who Masked: Participant, Investigator
Masking Description: Double-blinded parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a supplement to take daily for 4 weeks. The supplement contains a combination of a protein hydrolysate and beta-glucan (Wellmune®).
  Interventions: Dietary Supplement: Supplement containing a protein hydrolysate + beta glucan (Wellmune®)
- Control group (Placebo Comparator): The control group will consume a placebo supplement containing maltodextrin daily for 4 weeks.
  Interventions: Dietary Supplement: Placebo supplement containing maltodextron

INTERVENTIONS:
Dietary Supplement: Supplement containing a protein hydrolysate + beta glucan (Wellmune®) — Supplement taken daily for 4 weeks.
  Arms: Intervention group
Dietary Supplement: Placebo supplement containing maltodextron — Placebo supplement taken daily for 4 weeks.
  Arms: Control group

SUMMARY:
This is a randomized placebo-controlled study that aims to investigate the effect of a new maternal dietary supplement (protein hydrolysate/yeast beta-glucan combination) on mother and infant health.

DETAILED DESCRIPTION:
N=140 healthy pregnant multiparous females aged between 18-49 years will be recruited to the study during pregnancy or up to 4-weeks postpartum, n=70 consuming the supplement and n=70 consuming a placebo. Following successful recruitment and screening, researchers will complete 2 study visits at the participant's home. Visit 1 marks the start of the intervention period and Visit 2 marks the end of the intervention period.

Once the baseline data is completed (visit 1), the capsules will be provided to the mother. One capsule will be taken daily for 4 weeks. Capsules will be provided in convenient weekly tablet boxes. The return of used tablet boxes and counting missing capsules will monitor compliance. In addition, regular weekly contact will be maintained by phone and text message with participants to encourage adherence. In addition to the 2 study visits, all participants will receive an individual consultation with a lactation consultant to ensure breastfeeding techniques are appropriate and not a confounding factor in the breastmilk supply.

Data collection will include:

Anthropometric measurements include weight, height/length, and circumferences. Questionnaires will be used to collect birth data, demographic, lifestyle, breastfeeding and infant behavior, socio-economic status, health history, and gut health information.

Dietary intakes will be assessed using an online 24-hour recall tool. Blood samples will be collected from mothers by a trained phlebotomist. A 5mL aliquot of breast milk will be collected from a full breast milk expression in the 24 hours prior to the research nurse visit using an electric breast pump. Mothers will record the volume of milk expressed and the remainder will be stored by the mother for the infant. for will use an electric breast pump for a full breast expression. The aliquot will be refrigerated until the research nurse visit.

Mothers will collect a fecal sample from themselves and a fecal and urine sample from their baby in the 24 hours prior to the visit and will be stored in the freezer until the research nurse visit.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18-49 years
* Multiparous with one previously breastfed child (defined as breastfed for greater than or equal to 3 months, does not need to be exclusively breastfed)
* Delivered term
* Woman free of breast or nipple infections
* Woman willing to avoid other galactagogues/breastmilk supply stimulants while on study
* Woman not taking medications that will affect lactation
* Woman is the established carer for the infant
* Infant has no baseline abnormality.

Exclusion Criteria:

* Less than 18 years old or older than 49 years (at time of recruitment)
* Smokers
* Individuals that are not free-living e.g. institutes where meals are prepared in bulk such as nursing homes, prisons etc.
* An inability to read, write or understand English
* Following a strict prescribed diet for any reason; insulin dependent diabetes, coeliac disease, Crohn's disease etc. as this may result in an altered gastrointestinal function.
* Mother or child has a milk protein allergy
* Covid-19 at very high-risk group (defined by HSE)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Expression of inflammatory cytokines in blood - TNF-alpha | 4 weeks
  The effect of the dietary supplement on TNF-alpha expression in blood collected from mothers will be measured using a gene expression assay of more than 200 genes (e.g., IL-1, IL-6, IL-8, TNF-a) at baseline and endpoint (week 4). TNF-alpha expression will be measured as Ct values and reported as relative quantities.
Expression of inflammatory cytokines in blood - IL-8 | 4 weeks
  The effect of the dietary supplement on IL-8 expression in blood collected from mothers will be measured using a gene expression assay of more than 200 genes (e.g., IL-1, IL-6, IL-8, TNF-a) at baseline and endpoint (week 4). IL-8 expression will be measured as Ct values and reported as relative quantities.

SECONDARY OUTCOMES:
Digestive health - SAGIS score | 4 weeks
  The effect of the dietary supplement on the digestive health of the mother will be measured using the Structured Assessment of Gastrointestinal Symptoms Scale (SAGIS) questionnaire at baseline and endpoint (4 weeks). SAGIS assesses gastrointestinal symptoms using a Likert scale 0-4 which is summed to give the SAGIS score.
Markers of metabolic health in blood - glucose | 4 weeks
  The effect of the dietary supplement on glucose concentrations (mmol/L) in blood collected from mothers will be measured using the HORIBA Pentra C400 at baseline and endpoint (week 4).
Markers of metabolic health in blood - insulin | 4 weeks
  The effect of the dietary supplement on insulin concentrations (mU/L) in blood collected from mothers will be measured using the HORIBA Pentra C400 at baseline and endpoint (week 4).
Markers of metabolic health in blood - triacylglycerol | 4 weeks
  The effect of the dietary supplement on triacylglycerol concentrations (mmol/L) in blood collected from mothers will be measured using the HORIBA Pentra C400 at baseline and endpoint (week 4).
Markers of metabolic health in blood - cholesterol | 4 weeks
  The effect of the dietary supplement on cholesterol concentrations (mmol/L) in blood collected from mothers will be measured using the HORIBA Pentra C400 at baseline and endpoint (week 4).
Secretory IgA in breastmilk | 4 weeks
  The effect of the dietary supplement on secretory IgA concentrations (ng/mL) in breastmilk collected from mothers will be measured using an ELISA at baseline and endpoint (week 4).
Breastmilk production volumn | 4 weeks
  The effect of the dietary supplement on breastmilk production will be measured by a full breast expression (mL) at baseline and endpoint (week 4).
Expression of inflammatory cytokines in blood | 4 weeks
  The effect of the dietary supplement on inflammatory cytokines in blood collected from mothers will be measured using a gene expression assay of more than 200 genes (e.g., IL-1, IL-6, IL-8, TNF-a) at baseline and endpoint (week 4).
Microbiota profile in feces | 4 weeks
  The effect of the dietary supplement on the gut microbiota profile of fecal samples collected from mothers and infants. Gut microbiota will be profiled using 16S rRNA sequencing and QIIME software at baseline and endpoint (week 4).
Microbiota profile in breastmilk | 4 weeks
  The effect of the dietary supplement on the gut microbiota profile of breastmilk samples collected from mothers. Microbiota will be profiled using 16S rRNA sequencing and QIIME software at baseline and endpoint (week 4).

CONTACTS AND LOCATIONS:
Overall Officials: Aifric O'Sullivan, PhD, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
At the start of the study each participant will have a study code assigned to them. All of the data from the trials will be stored using these unique study codes. A file will be set up which will be stored in a location separate to the study data. This file will contain a list which will link each participants contact details to the corresponding ID code. All stored information will be encrypted and protected by a password that only the researcher and PI will know.